CLINICAL TRIAL: NCT06790082
Title: FAPI PET in Pleural Mesothelioma: The Diagnostic Accuracy and Clinical Value of FAPI PET at Diagnosis, Primary Staging, and the Feasibility of FAPI PET for Response Evaluation
Brief Title: The Diagnostic Accuracy and Clinical Value of FAPI PET in Pleural Mesothelioma
Acronym: FAPI-PM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Morten Bentestuen, Principal Investigator, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EU CT: 2024-514301-62-00; 2024-514301-62-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-10; First posted 2025-01-23 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-01

CONDITIONS: Pleural Mesothelioma; Pleural Diseases; Cancer; FAPI; Fibroblast Activation Protein Inhibitor
Keywords: FAPI; 68Ga-FAPI-46; PET/CT; Pleural Mesothelioma; FDG PET/CT
MeSH Terms: conditions — Mesothelioma, Malignant; Pleural Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Suspected pleural mesothelioma (Experimental): Patients with suspected pleural mesotheliom undergo an additional study specific [68Ga]Ga-FAPI-46 PET/CT at primary staging.
  Interventions: Drug: [68Ga]Ga-FAPI-46 PET/CT

INTERVENTIONS:
Drug: [68Ga]Ga-FAPI-46 PET/CT — Patients with suspected pleural mesothelioma undergo FAPI PET/CT in addition to conventional imaging at primary staging.
  The subgroup of patients undergoing anticancer treatment will undergo an additional FAPI PET/CT and FDG PET/CT after completing 2-3 series of anticancer treatment.
  Other Names: [68Ga]Gallium - Fibroblast Activation Protein Inhibitor-46 Positron Emission Tomography / Computer Tomography

SUMMARY:
Seventy (N=70) patients with suspected pleural mesothelioma (PM) lesions referred to pleural biopsy will be recruited, and undergo an additional FAPI PET/CT at primary staging.

The FAPI PET/CT results will be compared to conventional imaging (including FDG PET/CT). The diagnostic accuracy will be determined with histopathology as reference standard.

For patients undergoing anticancer treatment (chemotherapy, immunotherapy, other treatment), an additional FAPI PET/CT and an additional FDG PET/CT will be conducted after the study subjects have completed 2-3 series of anticancer treatment. The feasabilitiy of FAPI PET/CT in response evaluation will be investigated.

All study specific analyzes will be blinded and will not influence the patient management / treatment.

DETAILED DESCRIPTION:
A new and promising PET tracer has been developed: Gallium-68 labelled fibroblast activation protein inhibitor (FAPI). FAPI binds to fibroblast activation protein (FAP), a type II transmembrane protein, which is expressed and upregulated in cancer associated fibroblasts. FAPI PET/CT has been superior to FDG PET/CT regarding tumor detection rate in multiple cancer entities. When evaluating the clinical value of FAPI PET/CT compared to conventional imaging, including FDG PET/CT, studies have shown that FAPI PET/CT led to a revised staging in up to 25-30% of cancer patients, and a revised treatment in up to 20-30% of patients. The clinical interest in FAPI extends beyond the use as a diagnostic tool, as the 68Ga-isotope can be replaced by a β-emitting isotope, e.g., 177-Lu or 90-Y, enabling radionuclide therapy of FAPI-avid cancers.

FAP-immunohistochemistry (FAP-IHC) studies in PM have shown promising results, and - as PM is of mesodermal origin, FAP-overexpression has been observed in the cancer cells themselves.

To date, only two clinical FAPI PET study in PM has been conducted. In these studies uptake values were significantly higher for FAPI PET compared to FDG PET regarding primary tumors and lymph node metastases. Moreover, FAPI PET/CT led to upstaging in some of the patients compared to FDG PET/CT.

Based on pathological studies, implementation of FAPI PET/CT could be particularly beneficial in sarcomatoid and biphasic PM subtypes, which are characterized by aggressive growth and a worse prognosis compared to the epithelioid subtypes, however, non-epithelioid subtypes are underrepresented in FAPI PET studies to date.

PM in most cases is diagnosed at advanced stages of the disease and surgery with pleurectomy/decortication is only indicated in select cases with localized disease (approx. 30% of patients with the epithelioid subtype). Therefore, most patients undergo palliative treatment with either chemotherapy, immunotherapy, or radiotherapy. Considering the inherent limitations and difficulties for CT based response evaluation tools in PM, experts argue that response assessment using FDG PET/CT, i.e., PET Response Evaluation Criteria in Solid Tumors (PERCIST), could be an even more sensitive tool in PM compared to anatomical imaging response tools.

To date, there are no studies evaluating the feasibility of FAPI PET for response assessment in PM.

The study is a prospective explorative study complying with the Standard for Reporting Diagnostic Accuracy (STARD) criteria where 70 patients with suspected PM are recruited.

An additional FAPI PET/CT will be performed as a study specific procedure at primary staging within 4 weeks of the primary staging FDG PET/CT and prior to the pleural biopsy. All included study subjects will undergo this additional primary staging FAPI PET/CT. Patients with benign histology will not receive any further study related procedures - unless they are re-recruited at a later time point. For the proportion of study subjects treated with chemotherapy or immunotherapy (anticancer treatment), as part of common clinical practice, additional study specific FAPI PET/CT and FDG PET/CT will be conducted after completing 2-3 series of anticancer treatment, that is 3 series of chemotherapy or 2 series of immunotherapy.

The study specific procedures will be conducted in addition to common clinical practice and will not interfere with or delay the routine diagnostic workup or treatment. The results of the study specific procedures will not be available to the patient or the treating physicians (blinded) and will not interfere with planned treatment/diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pleural lesions suspicious of pleural mesothelioma and referred to pleural biopsy.
* Undergone/undergoing FDG PET/CT as part of the diagnostic workup of a suspicious PM lesion.
* Considered physically and mentally able to participate in the research project.
* Understands the study subject information and able to consent to project participation.
* 18-years or older

Exclusion Criteria:

* Patients with an imminent need for surgery or in an emergency
* Known concurrent other malignancy with active treatment within the last 1 year; non-melanoma skin cancer and cervical cancer in situ are exempt.
* Pregnant or breastfeeding women.
* Fertile women (women of childbearing potential) who could - theoretically - be pregnant (i.e., unknown pregnancy status).

Fertile women will be tested for pregnancy (by urine humane choriogonadotropin (HCG) or serum HCG) within 48h before FAPI PET/CTs, both at primary staging and restaging. Study subjects can participate in the study if the pregnancy test is negative (i.e., not pregnant).

* Subjects unable to undergo PET/CT: e.g., weighing more than 180 kg (weight limit scanner), unable to fit within the imaging gantry, inability to remain still for the duration of the examination, or with known severe claustrophobia unresponsive to oral anxiolytics or severe fear of needles.
* Subjects with any medical condition or other circumstances that, in the opinion of the Investigator, would significantly decrease the reliability of data, achievement of study objectives or completing the study.
* History of allergic reactions / hypersensitivity attributed to [18F]FDG or FAPI-tracers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2037-04-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance | 2 years
  The diagnostic performance (sensitivity, specificity, positive predicative value, negative predicative value, and overall diagnostic accuracy - all parameters in %). in of FAPI PET compared to routine imaging modalities, including FDG PET/CT, in suspected PM lesions.

SECONDARY OUTCOMES:
Location biopsy | 2 years
  Calculate the proportion of patients where the location of the intended pleural biopsy is altered due to FAPI PET/CT replacing FDG PET/CT.
Staging | 2 years
  Compare the cancer stage (IASCL 9th edition TNM-classification) as determined by FAPI PET/CT compared to conventional imaging (including FDG PET/CT) at primary staging.
Patient Management | 2 years
  Calculate the proportion of patients with suspected PM lesion with a change in treatment following the -hypothetical - addition of FAPI PET/CT at primary staging.
Uptake Values | 2.5 years
  Investigate the FAPI PET uptake parameters in suspicious PM lesions (primary tumor), regional lymph nodes, and distant metastases, and in benign lesions. Correlate FAPI uptake parameters in different PM sutypes.
Changes uptake parameters due to anticancer treatment | 2.5 years
  Calculate changes in FAPI PET uptake parameters - from before to after 2-3 series of anticancer treatment. Changes will be presented as ratios and in %.
Correlate immunohistochemistry | 5 years
  Correlate the FAPI PET SUV to FAP targeting immunohistochemistry of biological material.
Incidental findings | 3 years
  Seek supplementary information in medical records, biochemistry, pathology, or other imaging modalities for a final diagnosis/condition in cases of unexpected FAPI PET/CT findings.
Safety Evaluation FAPI-injection | 2.5 years
  Report Incidence Treatment-Emergent Adverse Events
Overall survival | 10 years
  A 10 year follow up of included patients will be conducted to determine overall survival (OS) in days from diagnosis, correlated to FAPI PET/CT results.
Recurrence/Progression Free Survival | 10 years
  A 10 year follow up of included patients will be conducted to determine Recurrence Free Survival (RFS) and Progression Free Survival (PFS) in days from diagnosis, correlated to FAPI PET/CT results.
Response evaluation | 10 years
  Compare conventional CT-based response assessment (mRECIST/iRECIST) to PET based response assessment (PERCIST, and other FDG and FAPI PET derived data) to the clinical outcome, i.e., OS, RFS/PFS.
Interobserver reliability | 5 years
  Conduct an interobserver study of FAPI PET/CTs. Cohens Kappa d will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Zacho, MD, DMSc, Study Director — Clinical Professor dept. of Nuclear Medicine, Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Region North Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guglielmo P, Crivellaro C, Castello A, Della Corte CM, Pagano M, Marchesi S, Occhipinti M, Zucali PA, Evangelista L. Emerging Radiopharmaceuticals in Pet Imaging for Mesothelioma: A Review of [18F]FDG Alternatives. Mol Diagn Ther. 2025 Jan;29(1):55-66. doi: 10.1007/s40291-024-00756-4. Epub 2024 Nov 8. PMID 39514167
- [Background] Guzel Y, Komek H, Can C, Kaplan I, Kepenek F, Ebinc S, Buyukdeniz MP, Gundogan C, Oruc Z. Comparison of the role of 18 F-fluorodeoxyglucose PET/computed tomography and 68 Ga-labeled FAP inhibitor-04 PET/CT in patients with malignant mesothelioma. Nucl Med Commun. 2023 Jul 1;44(7):631-639. doi: 10.1097/MNM.0000000000001702. Epub 2023 Apr 28. PMID 37114422
- [Background] Kessler L, Schwaning F, Metzenmacher M, Pabst K, Siveke J, Trajkovic-Arsic M, Schaarschmidt B, Wiesweg M, Aigner C, Plones T, Darwiche K, Bolukbas S, Stuschke M, Umutlu L, Nader M, Theegarten D, Hamacher R, Eberhardt WEE, Schuler M, Herrmann K, Fendler WP, Hautzel H. Fibroblast Activation Protein-Directed Imaging Outperforms 18F-FDG PET/CT in Malignant Mesothelioma: A Prospective, Single-Center, Observational Trial. J Nucl Med. 2024 Aug 1;65(8):1188-1193. doi: 10.2967/jnumed.124.267473. PMID 38960716